CLINICAL TRIAL: NCT05623371
Title: Leading Well-being and the Psychosocial Working Environment - A Cluster-randomized Waitlist Controlled Trial of a Training Program for Middle Managers in a Danish Healthcare Setting
Brief Title: Leading Well-being and the Psychosocial Working Environment - A Cluster-randomized Waitlist Controlled Trial
Acronym: Matterhorn
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Central Denmark Region (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Matterhorn
Record Dates: First submitted 2022-10-12; First posted 2022-11-21 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-09

CONDITIONS: Stress; Well-being; Burn Out
Keywords: Manager training; stress; well-being; the psychosocial working environment
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: Cluster, randomized waitlist controlled trial. The treatment group receives the intervention in 2023, and the control group receives it in 2024.
Who Masked: Outcomes Assessor
Masking Description: As the design is a waitlist controlled trial, the participants, the consultans and the some of the involved researchers will know what individuals received the intervention in 2023 (i.e. the treatment group), and 2024 (i.e. the control group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Leadership training comprising 5 modules and group exercises
  Interventions: Behavioral: Training leaders in leading well-being and the psychosocial working environment
- Control group (Other): Active control group receiving the offer of a webinar and written material
  Interventions: Behavioral: The offer of a webinar and written material

INTERVENTIONS:
Behavioral: Training leaders in leading well-being and the psychosocial working environment — The intervention comprises five training modules with practice in small groups in between. Training will take place over 5 months. The training will be received in groups of 20 and the training will be facilitated by 2 facilitators. Central themes of the training are:
  1. Self-care and well-being of the manager and how to cope with stress as a manager.
  2. Employee well-being and reducing risk-factors in the psychosocial working environment of employee mental health problems
  3. Enhancing protective factors social social support and a healthy team climate
  4. Responding to employees at risk and how to handle difficult conversations and procedures on return to work
  5. Managing well-being in employees during organizational change and final reflections
  The training will comprise video material and in person training of competencies and behaviors in group settings.
  The waitlist control group will receive an offer of a webinar and written information.
  Arms: Treatment group
Behavioral: The offer of a webinar and written material — The offer of a webinar plus written material
  Arms: Control group

SUMMARY:
The design comprises a cluster, randomized waitlist controlled design. The goal of the study is to prevent stress and burnout in middle managers and employees in a hospital setting. The study population is middle managers in a hospital setting.

The intervention comprises five training modules with practice in small groups in between. Training will take place over 5 months. The training will be received in groups of 20 middle managers and the training will be facilitated by 2 facilitators. Themes of training are inspired by the concept of Health Oriented Leadership which takes into account that the well-being of managers is important for the well-being of employees. Central themes of the training are: 1) Self-care and well-being of the manager and how to cope with stress as a manager. 2) Employee well-being and reducing risk-factors in the psychosocial working environment of employee mental health problems. 3) Enhancing protective factors social social support and a healthy team climate. 4) Responding to employees at risk and how to handle difficult conversations and procedures on return to work. 5) Managing well-being in employees during changes and pressure.

In order to establish commitment for the waitlist control group, the control group will receive an offer of a webinar and some written information.

Middle managers in both intervention arms will receive a questionnaire at baseline, after the intervention and at 6 months follow-up. The intervention group will also receive a short questionnaire after each training.

The following expectations are hypothesized:

The training will improve self-care and perceived staff-care in middle managers and employees in the intervention group when compared to the control group

The training will improve psychological outcomes of stress, well-being, exhaustion and psychological symptoms among middle managers and employees in the intervention group when compared to the control group

The training will improve the perceived psychosocial working environment (PSWE) among middle managers and employees in the intervention group when compared to the control group

The training will reduce sickness absence and retention among middle managers and employees in the intervention group when compared to the control group

Middle managers who adhere more to the training will experience larger improvements in self-care, staff-care and mental outcomes

DETAILED DESCRIPTION:
The design comprises a two-armed cluster, randomized waitlist controlled design. The goal of the study is to prevent stress and burnout in middle managers and employees in a hospital setting. The study population is middle managers in a hospital setting. These managers are randomized by unit and stratified on number of managers enrolled from each unit to obtain equal numbers in each arm.

The intervention comprises five training modules with practice in small groups in between. Training will take place over 5 months. The training will be received in groups of 20 middle managers and the training will be facilitated by 2 facilitators. Themes of training are inspired by the concept of Health Oriented Leadership which takes into account that the well-being of middle managers is important for the well-being of employees. Central themes of the training are: 1) Self-care and well-being of the manager and how to cope with stress as a manager. 2) Employee well-being and reducing risk-factors in the psychosocial working environment of employee mental health problems. 3) Enhancing protective factors social social support and a healthy team climate. 4) Responding to employees at risk and how to handle difficult conversations and procedures on return to work. 5) Managing well-being in employees during changes and pressure.

In order to establish commitment for the waitlist control group, the control group will receive an offer of a webinar and some written information.

Middle managers in both intervention arms will receive a questionnaire at baseline, after the intervention and at 6 months follow-up. The intervention group will also receive a short questionnaire after each training.

The following expectations are hypothesized:

The training will improve self-care and perceived staff-care in middle managers and in employees in the intervention group when compared to the control group

The training will improve psychological outcomes of stress, well-being, exhaustion and psychological symptoms among middle managers and employees in the intervention group when compared to the control group

The training will improve the perceived psychosocial working environment (PSWE) among middle managers and employees in the intervention group when compared to the control group

The training will reduce sickness absence and retention among middle managers and employees in the intervention group when compared to the control group

Middle managers who adhere more to the training will experience larger improvements in self-care, staff-care and mental outcomes

ELIGIBILITY:
Inclusion Criteria:

* Included managers are middle managers in hospitals in the Danish Central Region
* Included managers must be directly responsible for employees
* Included managers must be responsible for yearly assesment talks

Exclusion Criteria:

* If the above is not true, based on the data collected when the manager signed up for the study, the manager is not included in the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-05-15 (Actual); Primary Completion 2024-01-08 (Estimated); Study Completion 2024-01-08 (Estimated)

PRIMARY OUTCOMES:
Change in perceived selfcare in middle managers and employees | Baseline, post training (6 months follow-up) and 12 months follow-up
  Measured with 16 items using an adapted version of the selfcare scale from The Health-Oriented Leadership questionnaire (Franke et al. 2014). Items are scored using a 5 point Likert scale ranging from 1 (a very low degree) to 5 (a very high degree) indicating to which extent they practice selfcare in relation to their work life
Change in perceived Staffcare in middle managers and employees | Baseline, post training (6 months follow-up) and 12 months follow-up
  Measured with 18 items using an adapted version of the staffcare scale from The Health-Oriented Leadership questionnaire (Franke et al. 2014). Items are scored using a 5 point Likert scale ranging from 1 (a very low degree) to 5 (a very high degree) indicating to which extent they practice selfcare in relation to their work life.
Change in perceived stress in middle managers and employees | Baseline, post training (6 months follow-up) and 12 months follow-up
  Measured with the Danish consensus version of the Perceived Stress Scale 10 (Eskildsen et al. 2015). The scale comprises 10 items measured on a five point likert scale ranging from 0 (never) to 4 (very ofte). A higher score indicates higher stress levels.
Change in burnout in middle managers and employees | Baseline, post training (6 months follow-up) and 12 months follow-up
  Measured with the Copenhagen Burnout Inventory. 19 Items are answered on a 6-point likert scale ranging from 0 (never) to 5 (always). The CBI understands the core components of burnout as fatigue and exhaustion.
Registered sickness absence in middle managers and employees | 12 months
  Measured with registered sickness absence from the business Intelligence department at the Central Denmark Region administration of sick-leave
Change in job satisfaction in middle managers and employees | Baseline, post training (6 months follow-up) and 12 months follow-up
  Measured with the Danish Psychosocial Questionnaire (Clausen et al. 2019), the job satisfaction item is scored on scale ranging from 0 (very unsatisfied) to 10 (very satisfied)

SECONDARY OUTCOMES:
Change in Well-being among middle managers and employees | Baseline, post training (6 months follow-up) and 12 months follow-up
  Measured with the WHO-5 well-being index (Bech et al. 2003). Items are answered on a 6 point Likert scale from 0 (at no time point) till 5 (all the time). The scale ranges from 0-100 where a higher score indicates higher well-being
Change in the perceived psychosocial working environment in middle managers and employees | Baseline, post training (6 months follow-up) and 12 months follow-up
  Measured with one item from the Danish Psychosocial Questionnaire (Clausen et al 2019).The job satisfaction item is scored on scale ranging from 0 (very unsatisfied) to 10 (very satisfied)
Change in perceive leadership quality among employees | Baseline, post training (6 months follow-up) and 12 months follow-up
  Measured with four items from the Danish Psychosocial Questionnaire (Clausen et al 2019). Items were scored on a 5 point Likert scale ranging from 1 (to a very high extent) to 5 (to a very low extent)
Change in central aspects of the psychosocial work environment among employees in employees | Baseline, post training (6 months follow-up) and 12 months follow-up
  Measured with the Danish Psychosocial Questionnaire (Clausen et al 2019). Addresses areas as influence, recognition, possibilities to conduct work tasks, predictability, recognition, social support from manager and colleagues quantitative and emotional demands, justice, work-life balance.
  Items are scored on a 5 point Likert scale ranging from 1 (to a very high extent) to 5 (to a very low extent)
Change in turnover intention among middle managers and employees | Baseline, post training (6 months follow-up) and 12 months follow-up
  Measured with a self-formulated single-item
Actual turnover among employees | 12 months
  Measured with registered sickness absence from the business Intelligence department at the Central Denmark Region administration of sick-leave
Change in perceived confidence among middle managers | Baseline, post training (6 months follow-up) and 12 months follow-up
  Modified version of items used in A New Online Mental Health Training Program for Workplace Managers: Pre-Post Pilot Study Assessing Feasibility, Usability, and Possible Effectiveness by Gayed et al. 2018
  Items were scored on a 5 point Likert scale ranging from 1 (to a very low degree) to 5 (to a very high degree)
Psychological saftety | Baseline, post training (6 months follow-up) and 12 months follow-up
  Measured five items from with scale by Edmonson 2018 items were scored on a scale from 1 (completely disagree) to 5 (completely agree) A higher score indicate a higher level of psychological safety
Psychosocial safety climate among employees | Baseline, post training (6 months follow-up) and 12 months follow-up
  Measured six items using an adapted version of the Psychosocial Safety Climate measure (PSC-12) items were scored on a scale from 1 (completely disagree) to 5 (completely agree)

OTHER OUTCOMES:
Questions on readiness among participating middle managers | 12 months
  Self-formulated process questions on readiness and adherence
Compliance with training programme among participating middle managers | 6 months
  Measured with administrative data on attendance at each module of the training program
Distress symptoms among middle managers and employees | 12 months
  Measured with Symptom Checklist, SCL-90-R
Change in sleep quality among middle managers and employees | Baseline, post training (6 months follow-up) and 12 months follow-up
  Two items from the Karolinska Sleep Questionnaire. Items were answered on a 5 point Likert scale ranging 1 (bad) to extremely good (5)
Change in knowledge on main topics among participating middle managers | Baseline, post training (6 months follow-up) and 12 months follow-up
  Self-formulated questions on degree of knowledge
Change in attitudes towards managing well-being among participating middle managers | Baseline, post training (6 months follow-up) and 12 months follow-up
  Self-formulated questions on attitude
Change in behavior aimed at managing well-being among participating middle managers | Baseline, post training (6 months follow-up) and 12 months follow-up
  Self-formulated questions on behavior
Change in Perceived quality of patient care among employees | Baseline, post training (6 months follow-up) and 12 months follow-up
  Self-formulated questions on perceived quality of patient care

CONTACTS AND LOCATIONS:
Overall Officials: Vita LP Dalgaard, Ph.D, Principal Investigator — Aarhus BSS, Aarhus University
Locations (1):
- Aarhus Universitet, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No
Due to data security regulation is it not possible to make individual participant data available to other researchers outside Aarhus University

REFERENCES:
- [Background] Andersen LL, Thorsen SV, Larsen M, Sundstrup E, Boot CR, Rugulies R. Work factors facilitating working beyond state pension age: Prospective cohort study with register follow-up. Scand J Work Environ Health. 2021 Jan 1;47(1):15-21. doi: 10.5271/sjweh.3904. Epub 2020 May 28. PMID 32463101
- [Background] Skakon J, Nielsen K, Borg V, Guzman J. Are leaders' well-being behaviours and style associated with the affective well-being of employees? A systematic review of three decades of research. Work and Stress - WORK STRESS. 2010;24:107-39.
- [Background] Petrie K, Gayed A, Bryan BT, Deady M, Madan I, Savic A, Wooldridge Z, Counson I, Calvo RA, Glozier N, Harvey SB. The importance of manager support for the mental health and well-being of ambulance personnel. PLoS One. 2018 May 23;13(5):e0197802. doi: 10.1371/journal.pone.0197802. eCollection 2018. PMID 29791510
- [Background] Harms PD, Credé M, Tynan M, Leon M, Jeung W. Leadership and stress: A meta-analytic review. The Leadership Quarterly. 2017;28(1):178-94
- [Background] Gayed A, Milligan-Saville JS, Nicholas J, Bryan BT, LaMontagne AD, Milner A, Madan I, Calvo RA, Christensen H, Mykletun A, Glozier N, Harvey SB. Effectiveness of training workplace managers to understand and support the mental health needs of employees: a systematic review and meta-analysis. Occup Environ Med. 2018 Jun;75(6):462-470. doi: 10.1136/oemed-2017-104789. Epub 2018 Mar 21. PMID 29563195
- [Background] Milligan-Saville JS, Tan L, Gayed A, Barnes C, Madan I, Dobson M, Bryant RA, Christensen H, Mykletun A, Harvey SB. Workplace mental health training for managers and its effect on sick leave in employees: a cluster randomised controlled trial. Lancet Psychiatry. 2017 Nov;4(11):850-858. doi: 10.1016/S2215-0366(17)30372-3. Epub 2017 Oct 12. PMID 29031935
- [Background] Taris TW, Nielsen K. Leadership in occupational health psychology. Work & Stress. 2019;33(2):105-6.
- [Background] Rugulies R. What is a psychosocial work environment? Scand J Work Environ Health. 2019 Jan 1;45(1):1-6. doi: 10.5271/sjweh.3792. No abstract available. PMID 30643919
- [Background] Harvey SB, Modini M, Joyce S, Milligan-Saville JS, Tan L, Mykletun A, Bryant RA, Christensen H, Mitchell PB. Can work make you mentally ill? A systematic meta-review of work-related risk factors for common mental health problems. Occup Environ Med. 2017 Mar;74(4):301-310. doi: 10.1136/oemed-2016-104015. Epub 2017 Jan 20. PMID 28108676
- [Background] Nieuwenhuijsen K, Verbeek JH, de Boer AG, Blonk RW, van Dijk FJ. Supervisory behaviour as a predictor of return to work in employees absent from work due to mental health problems. Occup Environ Med. 2004 Oct;61(10):817-23. doi: 10.1136/oem.2003.009688. PMID 15377767
- [Background] Ladegaard Y, Skakon J, Elrond AF, Netterstrom B. How do line managers experience and handle the return to work of employees on sick leave due to work-related stress? A one-year follow-up study. Disabil Rehabil. 2019 Jan;41(1):44-52. doi: 10.1080/09638288.2017.1370733. Epub 2017 Aug 28. PMID 28845715
- [Background] Bryan BT, Gayed A, Milligan-Saville JS, Madan I, Calvo RA, Glozier N, Harvey SB. Managers' response to mental health issues among their staff. Occup Med (Lond). 2018 Sep 13;68(7):464-468. doi: 10.1093/occmed/kqy103. PMID 30060150
- [Background] Tafvelin S, Hasson H, Nielsen K, Von Thiele Schwarz U. Integrating a transfer perspective into evaluations of leadership training. Leadership and Organization Development Journal. 2021;ahead-of-print.
- [Background] von Thiele Schwarz U, Nielsen K, Edwards K, Hasson H, Ipsen C, Savage C, Simonsen Abildgaard J, Richter A, Lornudd C, Mazzocato P, Reed JE. How to design, implement and evaluate organizational interventions for maximum impact: the Sigtuna Principles. Eur J Work Organ Psychol. 2020 Aug 26;30(3):415-427. doi: 10.1080/1359432X.2020.1803960. eCollection 2021. PMID 34518756
- [Background] Lacerenza CN, Reyes DL, Marlow SL, Joseph DL, Salas E. Leadership training design, delivery, and implementation: A meta-analysis. J Appl Psychol. 2017 Dec;102(12):1686-1718. doi: 10.1037/apl0000241. Epub 2017 Jul 27. PMID 28749153
- [Background] Nielsen K, Abildgaard JS. Organizational interventions: A research-based framework for the evaluation of both process and effects. Work & Stress. 2013;27:278-97.
- [Background] Franke, F., Felfe, J., and Pundt, A. (2014). The impact of health-oriented leadership on follower health: development and test of a new instrument measuring health-promoting leadership. German J. Hum. Resour. Manag. 28, 139-161. doi: 10.1177/239700221402800108
- [Background] Eskildsen A, Dalgaard VL, Nielsen KJ, Andersen JH, Zachariae R, Olsen LR, Jorgensen A, Christiansen DH. Cross-cultural adaptation and validation of the Danish consensus version of the 10-item Perceived Stress Scale. Scand J Work Environ Health. 2015 Sep 1;41(5):486-90. doi: 10.5271/sjweh.3510. Epub 2015 Jun 25. PMID 26111225
- [Background] Kristensen TS, Borritz M, Villadsen E, Christensen KB. The Copenhagen Burnout Inventory: a new tool for the assessment of burnout. Work Stress 2005;19:192-207.
- [Background] Clausen T, Madsen IE, Christensen KB, Bjorner JB, Poulsen OM, Maltesen T, Borg V, Rugulies R. The Danish Psychosocial Work Environment Questionnaire (DPQ): Development, content, reliability and validity. Scand J Work Environ Health. 2019 Jul 1;45(4):356-369. doi: 10.5271/sjweh.3793. Epub 2018 Dec 28. PMID 30592500
- [Background] Olsen LR, Mortensen EL, Bech P. The SCL-90 and SCL-90R versions validated by item response models in a Danish community sample. Acta Psychiatr Scand. 2004 Sep;110(3):225-9. doi: 10.1111/j.1600-0447.2004.00399.x. PMID 15283743
- [Background] Bech P, Olsen LR, Kjoller M, Rasmussen NK. Measuring well-being rather than the absence of distress symptoms: a comparison of the SF-36 Mental Health subscale and the WHO-Five Well-Being Scale. Int J Methods Psychiatr Res. 2003;12(2):85-91. doi: 10.1002/mpr.145. PMID 12830302
- [Derived] Dalgaard VL, Gayed A, Hansen AKL, Grytnes R, Nielsen K, Kirkegaard T, Uldall L, Ingerslev K, Skakon J, Jacobsen CB. A study protocol outlining the development and evaluation of a training program for frontline managers on leading well-being and the psychosocial work environment in Danish hospital settings - a cluster randomized waitlist controlled trial. BMC Public Health. 2023 May 10;23(1):848. doi: 10.1186/s12889-023-15728-2. PMID 37165331